CLINICAL TRIAL: NCT03732872
Title: Risk Assessment of Malignant Transformation in Oral Submucous Fibrosis Using Epithelial Mesenchymal Transition (EMT) Signatures in Tissue Samples and Saliva
Brief Title: Epithelial Mesenchymal Transition Markers in OSMF
Status: Completed | Type: Observational
Sponsor: The Oxford Dental College, Hospital and Research Center, Bangalore, India (Other)
Collaborators: Credora Life Sciences, India (Unknown)
Responsible Party: Principal Investigator, Dr. Shesha Prasad, Senior lecturer, The Oxford Dental College, Hospital and Research Center, Bangalore, India
Other Study IDs: Oxford DC
Record Dates: First submitted 2018-10-27; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Oral Submucous Fibrosis
Keywords: OSMF; EMT; miRNA 21; vimentin; e-cadherin
MeSH Terms: conditions — Oral Submucous Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. Patient tissue samples taken in biopsy from all three groups
  2. Saliva samples taken from all three groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with habits and having OSMF: Patients who had history of arecanut chewing habit in any form and composition and who were not undergone any treatment for their current condition i.e, OSMF
  Interventions: Diagnostic Test: Biopsy tissue analysis; Diagnostic Test: Saliva analysis
- Patients with habits and had no clinical symptoms of OSMF: Patients who had history of arecanut chewing habit in any form and composition and had no symptoms of OSMF clinically
  Interventions: Diagnostic Test: Biopsy tissue analysis; Diagnostic Test: Saliva analysis
- Healthy human volunteers: patients who reported no history of areacnut chewing habits and had no clinical symptoms of OSMF
  Interventions: Diagnostic Test: Biopsy tissue analysis; Diagnostic Test: Saliva analysis

INTERVENTIONS:
Diagnostic Test: Biopsy tissue analysis — biopsy samples for IHC staining and PCR
Diagnostic Test: Saliva analysis — Saliva samples for miRNA 21 expression analysis

SUMMARY:
Oral Sub mucous Fibrosis (OSMF) is essentially an imbalance between collagen metabolism and wound healing mechanism induced by arecanut chewing habit. Clinically the disease progresses in stages with patients presenting with burning sensation, intolerance to spicy food, vesicles particularly on the palate, ulceration and dryness of the mouth , fibrosis of the oral mucosa, leading to lips, tongue, and palate rigidity and finally trismus. As the disease is progressively debilitating and has potential to turn in to malignant cancer a study was designed to assess if there any tissue or saliva markers that can be assessed for early diagnosis and indicate malignant transformation if any.

Participants who had OSMF and habit history, patients without OSMF but habit history formed the case group where as normal patients without OSMF and no habit history were in control group. Eligible candidates who consented to participate in study were subjected to biopsy procedure and also their saliva samples were collected. Biopsy samples were subjected to immunohistochemistry (IHC) and polymerase chain reaction (PCR) to assess the EMT markers like vimentin, e-cadherin and collagen IV. miRNA copies were extracted from saliva and were subjected RT-PCR.

Research question was:

1. Is EMT a positive signature in OSMF.
2. Does histopathological grading and dysplasia in OSMF have any correlation with EMT.
3. Can aberrant EMT markers be a reliable indicator for risk assessment of early malignant transformation.
4. Can expression of mi RNA 21 in saliva predict the disease severity and more importantly assess risk of early malignant transformation in OSMF.

DETAILED DESCRIPTION:
Epithelial-mesenchymal transition (EMT) describes the process whereby cells shed their epithelial properties and adopt a more mesenchymal and invasive phenotype. A continuous molecular cross talk between epithelial and mesenchymal cells is required during embryonic development (epithelial mesenchymal transition) and probably plays an important role in pathologic process like wound healing and tumour progression. The development of carcinomas is due to the genetic changes within the target epithelium. As there is conversion of normal epithelium to potentially malignant and to squamous cell carcinoma, the stroma also changes from normal to activated or tumor associated called as the stromal reaction. 10 EMT can generate mesenchymal cells that express α-smooth muscle actin (αSMA), as seen in myofibroblasts. It is, however, unclear whether functional myofibroblasts seen in fibrosis or cancer derived from epithelial or endothelial cells

Hence EMT markers in OSMF were assessed in this study. the following markers chosen as:

1. miRNA-21 regulates cell proliferation, apoptosis and the epithelial to mesenchymal transition during neoplastic progression and is up regulated in a variety of cancers.An increased expression of miRNA-21 is seen in myofibroblasts.12 Since we know the role of myofibroblasts in OSMF, salivary expression of mi RNA- 21 was included as marker.
2. Type IV collagen has the unique feature of self-associating through intramolecular covalent bonds, providing barrier and mechanical strength properties to basement membranes.The increased collagen deposition in OSMF involves numerous fibroblasts that are converted to myofibroblasts found in histologic sections of tissue specimens. an altered micro environment or stroma such as persistent myofibroblasts has been shown to result in tumorigenesis and tumor progression
3. Cadherins are a class of type-1 trans-membrane proteins known for its calcium-dependent cell-cell adhesion property. E-cadherins are members of this protein family found in epithelial cells which serve important roles in cell adhesion by ensuring that cells within tissues are bound together. The loss of E-cadherin function or expression has been implicated in cancer progression and metastasis.E-cadherin expression in the head and neck epithelium is essential for the morphogenesis and homeostasis of epithelial tissues. The cadherin-mediated cell-cell contacts are required for the anchorage-dependent growth of epithelial cells.

   Hence lower expression of E- cadherin is a sign of loss of epithelial integrity
4. The intermediate filament protein vimentin is involved in the regulation of cell behavior, morphology, and mechanical properties. Vimentin is a EMT marker expressed in connective tissue. Expression of vimentin in epithelium is a positive signature of EMT, and its evaluation in OSMF can unveil the importance of EMT signature in oral fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who had history of arecanut chewing habit with clinical manifestations of OSMF.
* Patients who had arecanut chewing habit history of more than 1 year and had no clinical symptoms of OSMF.
* Healthy human volunteers who are indicated for extraction of tooth and had no clinical features of OSMF and had no habit history

Exclusion Criteria:

* Patients who had bleeding disorders
* patients who are diagnosed with salivary gland disorders that can alter salivary flow or composition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were selected from outpatient department of Dental College OPD
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Expression of E-cadherin levels in all the groups in IHC | 10 days from sample collection
  For IHC: The criteria used to define E-cadherin positive cells was brown staining in cell membrane of epithelial cells; the percentage of positively stained cells were scored as -
  Percentage of POSITIVE CELLS SCORE No cells 0 ≤ 10% 1 11% -50 % 2 51%-80% 3
  ≥81% 4
  Staining Intensity was also assessed in comparison with the positive control tissue and scored accordingly
  INTENSITY SCORE Negative 0 Weak 1 Moderate 2 Strong 3
Change in Expression of vimentin levels in all the groups in IHC | 10 days from sample collection
  vimentin positive cells was brown staining in cytoplasm of epithelial cells; the percentage of positively stained cells were scored as -
  Percentage of POSITIVE CELLS SCORE No cells 0 ≤ 10% 1 11% -50 % 2 51%-80% 3
  ≥81% 4
  Staining Intensity was also assessed in comparison with the positive control tissue and scored accordingly
  INTENSITY SCORE Negative 0 Weak 1 Moderate 2 Strong 3
Change in Expression of collagen IV levels in all the groups in IHC | 10 days from sample collection
  collagen IV positive cells was brown staining in basement membrane cells; the percentage of positively stained cells were scored as -
  Percentage of POSITIVE CELLS SCORE No cells 0 ≤ 10% 1 11% -50 % 2 51%-80% 3
  ≥81% 4
  Staining Intensity was also assessed in comparison with the positive control tissue and scored accordingly
  INTENSITY SCORE Negative 0 Weak 1 Moderate 2 Strong 3
Change in Expression of miRNA 21 in all three groups using Real Time-PCR | 10 days from sample collection
  Considering the expression of miRNA21 in normal sample (N) as 1, the expression of all the samples were calculated The formula used is: number of copies = (amount * 6.022x1023) / (length * 1x109 * 650)
CHange in E cadherin levels in PCR | 20 days after sample collection
  After extraction of DNA from biopsy samples the primers for E-cadherin were designed using Primer Express software, synthesized and HPLC purified for real time PCR for quantification.
Change in vimentin levels in PCR | 20 days after sample collection
  After extraction of DNA from the biopsy samples the primers for Vimentin were designed using Primer Express software, synthesized and HPLC purified for real time PCR for quantification

SECONDARY OUTCOMES:
Change in e-cadherin expression with respect to disease category clinically in OSMF patients with habits | 15 days from sample collection
  E cadherin level in tissue samples with respect to different Clinical expression of disease according to Kerr et al classification system.
Change in e-cadherin expression with respect to disease category histologically in OSMF patients with habits | 15 days from sample collection
  E cadherin level in tissue samples with respect to different Clinical expression of disease according to Kanna and Andrade et al classification system.
Change in vimentin expression with respect to disease category clinically in OSMF patients with habits | 15 days from sample collection
  Vimentin level in tissue samples with respect to different Clinical expression according to Kerr et al classification system.
Change in vimentin expression with respect to disease category histologically in OSMF patients with habits | 15 days from sample collection
  Vimentin level in tissue samples with respect to different histological expression according to Khanna and Andrade classification system.
Change in collagen IV expression with respect to disease category clinically in OSMF patients with habits | 15 days from sample collection
  Collagen-IV level in tissue samples with respect to different Clinical expression category according to Kerr et al classification system.
Change in collagen IV expression with respect to disease category hstologically in OSMF patients with habits | 15 days from sample collection
  Collagen-IV level in tissue samples with respect to different histological expression according to Khanna and Andred et al classification system.
Change in mi RNA 21 expression with respect to disease category clinically in OSMF patients with habits | 15 days from sample collection
  miRNA 21 level in saliva samples with respect to different Clinical expression of OSMF according to Kerr et al classification system.
Change in mi RNA 21 expression with respect to disease category histologically in OSMF patients with habits | 15 days from sample collection
  miRNA 21 level in saliva samples with respect to different histological expression according to Khanna and Andred et al classification system.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Li YX, Yang X, Jiang L, Zhou ZJ, Zhu YQ. Progress risk assessment of oral premalignant lesions with saliva miRNA analysis. BMC Cancer. 2013 Mar 19;13:129. doi: 10.1186/1471-2407-13-129. PMID 23510112
- [Background] Sawant SS, Vaidya Mm, Chaukar DA, Alam H, Dmello C, Gangadaran P, Kannan S, Kane S, Dange PP, Dey N, Ranganathan K, D'Cruz AK. Clinical significance of aberrant vimentin expression in oral premalignant lesions and carcinomas. Oral Dis. 2014 Jul;20(5):453-65. doi: 10.1111/odi.12151. Epub 2013 Jul 19. PMID 23865921
- [Background] Pinto GA, Vassallo J, Andrade LA, Magna LA. Immunohistochemical study of basement membrane collagen IV in uterine cervix carcinoma. Sao Paulo Med J. 1998 Nov-Dec;116(6):1846-51. doi: 10.1590/s1516-31801998000600004. PMID 10349192